CLINICAL TRIAL: NCT06900257
Title: Evaluation of Fetal Cardiac Functions in Fasting Pregnant Women
Brief Title: Fetal Cardiac Functions in Fasting Pregnant Women
Status: Enrolling by invitation | Type: Observational
Sponsor: Sanliurfa Education and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: ŞEAH/fasting card
Record Dates: First submitted 2025-03-23; First posted 2025-03-28 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Fasting Pregnant Women
Keywords: Fasting; Pregnancy; Fetal echocardiography; Fetal health
MeSH Terms: conditions — Fasting | interventions — Pregnancy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Singleton uncomplicated pregnancies with at least 10 days of fasting.
  Interventions: Procedure: Pregnant women who present for routine antenatal follow-up between 24-34 weeks of gestation.
- The control group will consist of healthy pregnant women who do not fast, with singleton uncomplicat
  Interventions: Procedure: Pregnant women who present for routine antenatal follow-up between 24-34 weeks of gestation.

INTERVENTIONS:
Procedure: Pregnant women who present for routine antenatal follow-up between 24-34 weeks of gestation. — All singleton uncomplicated pregnancies that present to our hospital for routine antenatal follow-up between 24-34 weeks of gestation will be included in this study.

SUMMARY:
In this study, we aimed to evaluate fetal cardiac functions after a fasting period of at least 10 days. The purpose of this study was to determine the unexpected effects of fasting on fetal cardiac functions.

DETAILED DESCRIPTION:
Pregnancies at 24-34 weeks of gestation who present to our hospital for routine antenatal follow-up will be evaluated. As the study group, singleton uncomplicated pregnancies with at least 10 days of fasting will be assessed. All ultrasonographic examinations will be conducted within the last 2 hours of the fasting period. The control group will consist of healthy pregnant women who do not fast, with singleton uncomplicated pregnancies between 24-34 weeks, matched for age, parity, and gestational age.

ELIGIBILITY:
Inclusion Criteria:

* Singleton, uncomplicated pregnancies that have been fasting for at least the last 10 days
* Present for routine antenatal follow-up between 24-34 weeks of gestation

Exclusion Criteria:

* Multiple pregnancy
* Premature rupture of membranes
* Chorioamnionitis
* Placental abruption
* Severe fetal growth restriction
* Congenital fetal anomalies
* Preeclampsia
* Oligohydramnios
* Maternal diabetes -Conditions where fasting is contraindicated for the mother. -

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Singleton uncomplicated pregnancies that present for routine antenatal follow-up between 24-34 weeks of gestation.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Singleton uncomplicated pregnancies with at least 10 days of fasting. | Fetal echocardiographic findings after at least 10 days of fasting.

CONTACTS AND LOCATIONS:
Locations (1):
- Sanliurfa Education and Research Hospital, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No